CLINICAL TRIAL: NCT06265935
Title: The Effect of Diaphragmatic Breathing Exercise on Fatigue and Quality of Life in Pregnant Women With Gestational Diabetes
Brief Title: Effect of Diaphragmatic Breathing Exercise on Fatigue and Quality of Life in Pregnant Women With Gestational Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Neslihan Atli, midwife, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ataturk Unıversıty - Neslihan
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Pregnancy in Diabetic; Fatigue; Quality of Life
MeSH Terms: conditions — Pregnancy in Diabetics; Fatigue | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomize
Who Masked: Participant
Masking Description: The sample size was calculated as 60 pregnant women by performing GPower analysis, taking into account the tests to be used to calculate the minimum sample size to be included in the study. The sampling will include a total of 60 primiparous pregnant women, including 30 pregnant women diagnosed with gestational diabetes who meet the inclusion criteria for the study, who agree to participate in the study, and 30 pregnant women diagnosed with gestational diabetes who are applied diaphragmatic breathing exercise and who are not applied diaphragmatic breathing exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Breathing exercise will be explained to the pregnant woman, taught and applied for 5 minutes. When doing the diaphragmatic breathing exercise, you will be told to take chest breaths after 4-5 diaphragmatic breaths to prevent hyperventilation. Feedback will be received, questions will be answered, a training brochure will be given and the program will be completed. Pregnant women will be asked to bring the questionnaire with them to their follow-up in two weeks. The Visual Similarity Scale for Fatigue and the SF-36 Quality of Life Scale will be refilled. How he did the exercise, whether he felt any effects and his satisfaction will be questioned. Your questions will be answered. You will be notified that you need to come for a check-up again in two weeks. Visual Similarity Scale for Fatigue and SF-36 Quality of Life Scale will be completed.
  Interventions: Behavioral: Experimental Group
- Control Group (No Intervention): No treatment will be performed on the participants in the control group, and they will be asked not to engage in regular physical activity or sports for 4 weeks and not to make any changes in their living habits.
  Pregnant women will be asked to bring the survey form with them at the follow-up visits two weeks later. The Visual Similarity Scale for Fatigue and the SF-36 Quality of Life Scale will be refilled. You will be notified that you need to come for a check-up again in two weeks. At the follow-up after the fourth week, the Visual Similarity Scale for Fatigue and the SF-36 Quality of Life Scale will be filled out again. At the end of thirty days, the program will be completed and the forms will be filled.

INTERVENTIONS:
Behavioral: Experimental Group — It will be carried out as a randomized controlled experimental design to determine the fatigue and quality of life of pregnant women with gestational diabetes.
  Other Names: Control Group
  Arms: Experimental Group

SUMMARY:
Gestational diabetes mellitus (GDM) is one of the most common medical complications of pregnancy. GDM, which is in the high-risk pregnancy category, causes fatigue during pregnancy due to both hormonal changes and pregnancy complications (1). Fatigue is a general complaint that occurs in almost all physical and mental diseases. Fatigue also negatively affects an individual's well-being, daily performance, activities of daily living (ADLs) and relationships. Fatigue is one of the symptoms that, if not controlled, negatively affects the individual's daily living activities and quality of life (2). While breathing itself is a way of relaxation, it is also a part of all relaxation exercises and is an exercise that can be used in daily life. Breathing correctly and deeply is the first step in learning to relax. (3). It is important to identify fatigue, minimize it, plan daily living activities and improve quality of life in patients with GDM. This study will be conducted as a randomized controlled study to determine the fatigue and quality of life of diaphragmatic breathing exercises, one of the non-pharmacological methods, on pregnant women with gestational diabetes.

DETAILED DESCRIPTION:
It will be carried out as a randomized controlled experimental design to determine the fatigue and quality of life of pregnant women with gestational diabetes.

Material and method of the research:

Type of Study: This research is a randomized controlled study.

Research Questions/Hypotheses:

Hypothesis 0 (H0): Diaphragmatic breathing exercise has no effect on fatigue and quality of life in pregnant women with gestational diabetes.

Hypothesis 1 (H1): Diaphragmatic breathing exercise has an effect on fatigue and quality of life in pregnant women with gestational diabetes.

Location and Characteristics of the Research: The research will be conducted with pregnant women with gestational diabetes who applied to the gynecology outpatient clinic of Şanlıurfa Training and Research Hospital between 1 August 2023 and 1 August 2024 and who meet the inclusion criteria. This hospital was chosen due to its nature as a regional hospital and its density of pregnant women.

Population-sample of the research: The population of this research will consist of pregnant women with gestational diabetes who were followed in the gynecology outpatient clinic of Şanlıurfa Training and Research Hospital between 1 August 2023 and 1 August 2024. The sample size was calculated as 60 pregnant women by performing GPower analysis, taking into account the tests to be used to calculate the minimum sample size to be included in the study. The sampling will include a total of 60 primiparous pregnant women, including 30 pregnant women diagnosed with gestational diabetes, who meet the inclusion criteria for the study, who agree to participate in the study, who are subjected to diaphragmatic breathing exercise, and 30 pregnant women diagnosed with gestational diabetes, who are not applied diaphragmatic breathing exercise.

Data Collection Forms and Tools Pregnancy Identification Form: This form was prepared and developed by researchers based on the literature. It consists of questions aimed at determining the sociodemographic, medical and obstetric characteristics of pregnant women with gestational diabetes.

SF-36 Quality of Life Scale: SF-36 Quality of Life Scale is a self-assessment scale consisting of 36 questions and eight subscales, developed by Ware in 1987 to measure care outcomes in general, not specific to age, disease or treatment, and to examine health-related quality of life. . The second question of the scale includes the perception of change in health in the last 12 months, and the other questions are evaluated considering the last four weeks. The Physical and Mental Health Summary Score is obtained by weighting the scores of the questions containing the subscales of the SF-36 Quality of Life Scale. Total score calculation is not possible. The resulting summary scores and subscale scores are expressed as continuous variables ranging from 0 to 100. Zero indicates bad health, 100 indicates well-being. The scale has no cut-off point. The validity and reliability of the scale in Turkey was conducted by Pınar in 1995 on 50 cardiology, 50 hemodialysis and 80 diabetes mellitus patients. According to this; Regardless of patient groups, the test-retest reliability coefficient of the scale was found to be 0.94, and the Crohnbach's Alpha value, which indicates internal consistency, was 0.92 .

Visual Similarity Scale for Fatigue: It was developed by Lee et al. in 1990 to measure the level of fatigue in various populations, including healthy adults and those with chronic diseases. The validity and reliability study of the scale for our country was conducted by Yurtsever and Bedük in 2003. YİGBS consists of 18 items. Of these items, 13 items measure Fatigue and five items measure Energy sublevel. Each item of the scale has a 10 cm horizontal line with positive statements at one end and negative statements at the other end. People who fill out this scale are asked to mark the point that best reflects the emotion they feel when reading the statements on the scale. Then, the intersection point at the marked location is measured with a ruler separately for each question, and the measured length is determined as the score of that item and evaluated objectively. The highest score that can be obtained from the fatigue subscale is 130 and the lowest score is 0. The highest score that can be obtained from the energy subscale is 50 and the lowest score is 0. A high score from the Fatigue subscale and a low score from the Energy subscale indicate that the severity of fatigue is high.[2] Cronbach's Alpha internal consistency coefficient for the 13-item fatigue subscale of the scale was found to be 0.90, and for the five-item energy subscale was 0.74.

Diaphragmatic Breathing Exercise: In diaphragmatic breathing exercise; Individuals lie on their back with their legs flexed, a pillow under their head, and place their dominant hand on their abdomen and the other hand on their chest. While breathing slowly through the nose, they need to pay attention to the hand in the abdominal area and reduce the rib cage movement by increasing the abdominal movement. During inspiration, as air fills the lungs, the hand on the abdomen should rise up and the hand on the chest should not move too much. It makes participants feel relaxed and relaxed with breathing exercise.

Collection of Data Data will be obtained from pregnant women with gestational diabetes who apply to the gynecology clinic of Şanlıurfa Training and Research Hospital and meet the sample selection criteria. Before the application, an explanation will be given to the pregnant women about the purpose of the research, and if they volunteer, their verbal and written consent will be obtained through the "Informed Volunteer Consent Form". Information about pregnant women will be collected by the researcher.

Application of Research Pregnant women will be informed about the research and written and verbal permissions will be obtained.

Information about pregnant women will be recorded. Pregnant women with gestational diabetes, whose diagnosis of gestational diabetes has been decided by the physician and who have given consent to participate in the study, will be assigned to 2 groups by randomization method: experimental (diaphragmatic breathing exercise group) and control (diaphragmatic breathing exercise group).

The first evaluations of pregnant women in both groups will be carried out between 10:00-12:00, and the Pregnancy Identification Form, Visual Similarity Scale for Fatigue and SF-36 Quality of Life Scale will be applied to the pregnant women before the training.

Experimental Group: Breathing exercise will be explained to the pregnant woman in a way she can understand, will be taught and will be applied for 5 minutes. When doing the diaphragmatic breathing exercise, participants will be told to take one chest breath after 4-5 diaphragmatic breaths to avoid hyperventilation. The pregnant woman will be advised to close her eyes during exercise and concentrate on breathing and focus her attention in this direction. If there is tremors, sweating, restlessness, palpitations, numbness in the hands or lips, or uterine contraction, participants will be told to stop the exercise and rest for a few minutes. Pregnant women will be given a phone number they can reach at any time during the one-month program. Feedback will be received, questions will be answered, a training brochure will be given and the program will be completed.

During their follow-up two weeks later, pregnant women will be asked to bring the survey form with them. The Visual Similarity Scale for Fatigue and the SF-36 Quality of Life Scale will be completed again. How he did the exercise, whether he felt any effects, and his satisfaction will be questioned. Their questions will be answered. Participants will be informed that participants need to come for a re-check in two weeks.

The Visual Similarity Scale for Fatigue and the SF-36 Quality of Life Scale will be filled out again during the follow-up after the fourth week. At the end of 30 days, the program will be completed and the survey form will be received.

Control Group: No application will be performed with the participants in the control group, and these participants will be asked not to engage in regular physical activity or sports for 4 weeks and not to make any changes in their living habits.

During their follow-up two weeks later, pregnant women will be asked to bring the survey form with them. The Visual Similarity Scale for Fatigue and the SF-36 Quality of Life Scale will be completed again. Participants will be informed that participants need to come for a re-check in two weeks.

The Visual Similarity Scale for Fatigue and the SF-36 Quality of Life Scale will be filled out again during the follow-up after the fourth week. At the end of 30 days, the program will be completed and the forms will be filled.

Evaluation of Data Evaluation of the data obtained as a result of the research will be analyzed using the SPSS (Statistical Package For Social Sciences) 25.0 package program.

Limitation of the Study: It is limited to pregnant women who applied to Şanlıurfa Training and Research Hospital affiliated with Şanlıurfa Provincial Health Directorate.

Ethical and Legal Aspects of Research Permission will be obtained from Atatürk University Clinical Research Ethics Committee before data collection. Institutional permission will be obtained from Şanlıurfa Provincial Health Directorate. Before the application, pregnant women with gestational diabetes will be informed about the purpose of the research, and if they volunteer, their verbal and written consent will be obtained through the "Informed Volunteer Consent Form".

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 19-35,
* 24-28. During the pregnancy week,
* Being a single and live fetus,
* No reading and writing problems, no mental disabilities or communication problems.

Exclusion Criteria:

* Multiple pregnancy,
* Fetal congenital malformation,
* Having a diagnosed disease other than GDM
* There is a risk of miscarriage during pregnancy,

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 2 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
SF-36 Quality of Life Scale: | SF-36 Quality of Life Scale: Scale scores are expressed as a continuous variable ranging from 0 to 100. Zero indicates bad health, 100 indicates well-being.
  Experimental group

SECONDARY OUTCOMES:
Visual Similarity Scale for Fatigue | The highest score that can be obtained from the Fatigue subscale is 130 and the lowest score is 0. A high score from the Fatigue subscale and a low score from the Energy subscale indicate that the severity of fatigue is high.
  Control group

CONTACTS AND LOCATIONS:
Overall Officials: Hava Özkan, Study Chair — Ataturk University

IPD SHARING:
Plan to Share IPD: No